CLINICAL TRIAL: NCT05720052
Title: A Phase I/II Study to Evaluate the Safety and Efficacy of the MS-553 in Patients With Relapsed or Refractory B-cell Lymphoma
Brief Title: A Study of MS-553 in Patients With Relapsed or Refractory B-cell Lymphoma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The study is terminated due to major protocol revisions.
Sponsor: MingSight Pharmaceuticals, Inc (Industry)
Collaborators: Shenzhen MingSight Relin Pharmaceutical Co., Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-003-CN
Record Dates: First submitted 2023-01-11; First posted 2023-02-09 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-07

CONDITIONS: Relapsed or Refractory B-cell Lymphoma; Diffuse Large B-cell Lymphoma (DLBCL); Follicular Lymphoma (FL); Mantle Cell Lymphoma (MCL); Chronic Lymphocytic Leukemia (CLL); Small Lymphocytic Lymphoma (SLL); Marginal Zone Lymphoma (MZL)
MeSH Terms: conditions — Recurrence; Lymphoma, B-Cell; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, B-Cell, Marginal Zone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm (Experimental): dose exploration
  Interventions: Drug: MS-553

INTERVENTIONS:
Drug: MS-553 — MS-553 oral tablet BID x 28-days

SUMMARY:
This is a Phase I/II, single-arm, multicenter, open-label study which is divided into two portions: Phase I is dose escalation portion, in which subjects with relapsed or refractory B-cell lymphoma will be enrolled except malignant lymphoblastic lymphoma (LBL) and Burkitt lymphoma. After the RP2D is identified, Phase II of subjects with relapsed or refractory mantle cell lymphoma who previously received ≥ 2 and ≤ 4 different chemotherapy and/or targeted drug therapy will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* 1) Patients in Phase I study will be enrolled with refractory or relapsed B-cell non-Hodgkin lymphoma.
* 2) Patients enrolled in the phase I study failed two or more lines of treatment regimens; Patients with mantle cell lymphoma should also be patients with contraindications or failure of BTK inhibitor therapy.
* 3) Eastern Cooperative Oncology Group (ECOG) performance status score is 0~2.
* 4) Have life expectancy ≥ 3 months.
* 5) Major organ functions meet the following criteria:

  * In the absence of growth factor support therapy or blood transfusion in the last 14 days: absolute neutrophil count ≥1.5×109/L, hemoglobin ≥80 g/L, platelets ≥75×109/L (no platelet transfusion within 14 days); if accompanied with bone marrow invasion, neutrophils ≥1.0×109/L, platelets ≥50×109/L.
  * Biochemistry: Total bilirubin ≤1.5×ULN or ≤3.0×ULN in Gilbert's syndrome, AST or ALT ≤2.5×ULN, serum creatinine ≤1.5×ULN or calculated creatinine clearance ≥60 mL/min (Cockcroft-Gault formula).
  * Coagulation function: International normalized ratio (INR) and activated partial thrombin time ≤ 1.5 × ULN.

Exclusion Criteria:

* 1) Present or prior history of other malignancies (except cured carcinoma in situ of cervix and basal cell carcinoma of skin), unless there is radical treatment and no evidence of recurrence or metastasis within the last 2 years.
* 2) Lymphomas involved the central nervous system.
* 3) Patients with history of organ transplantation or allogeneic hematopoietic stem cell transplantation; patients who have received autologous hematopoietic stem cell transplantation or CAR-T treatment within the past 3 months,
* 4) Patients who are suitable and ready for autologous stem cell transplantation.
* 5) History of eye surgery or trauma within 3 months before the screening visit, history of serious eye infection or the most recent eye surgery within 4 weeks before the screening visit.
* 6) Has had active and uncontrolled autoimmune hemocytopenia, including autoimmune hemolytic anemia and idiopathic thrombocytopenic purpura.
* 7) Has had uncontrolled or significant cardiovascular diseases, including:
* 8) Women who are lactating or pregnant.
* 9) Women of child-bearing potential who do not agree to have two pregnancy tests prior to first dose (at least one of tests is serum pregnancy test) and the test result shall be negative.
* 10) Male patients who do not agree to the birth control measures.
* 11) Any conditions that in the opinion of the investigator considers inappropriate to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2023-02-06 (Actual); Primary Completion 2023-11-28 (Actual); Study Completion 2023-11-28 (Actual)

PRIMARY OUTCOMES:
Incidence of dose limiting toxicity (DLT) | First cycle (28 days)
Incidence and severity of adverse events | up to 24 months
To determine the MTD and RP2D of oral MS-553 in patients with BCL | about 8 months

SECONDARY OUTCOMES:
Objective response rate (ORR) | up to 24 months
Duration of response (DOR) | up to 24 months
progression-free survival (PFS) | up to 24 months
overall survival (OS) | up to 24 months
time to progression (TTR) | up to 24 months
disease control rate (DCR) | up to 24 months
Pharmacokinetics parameters: Cmax | within the first 2 cycles (56 days)
Pharmacokinetics parameters: Tmax | within the first 2 cycles (56 days)
Pharmacokinetics parameters: T1/2 | within the first 2 cycles (56 days)
Pharmacokinetics parameters: AUC0-12 | within the first 2 cycles (56 days)
Pharmacokinetics parameters: CL/F | within the first 2 cycles (56 days)

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Beijing, China